CLINICAL TRIAL: NCT05657119
Title: Family Safety Net: Developing an Upstream Suicide Prevention Approach to Encourage Safe Firearm Storage in Rural and Remote
Brief Title: Family Safety Net - Aim 3: Randomized Control Trial
Acronym: FSN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Maniilaq Association (Unknown)
Responsible Party: Principal Investigator, Lisa Wexler, Professor of Social Work, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00225431
Record Dates: First submitted 2022-12-01; First posted 2022-12-20 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Suicide; Accidental Injuries; Firearm Injury
Keywords: Motivational Interviewing; Suicide Prevention; Alaska Native; Firearm Storage; Family Engagement
MeSH Terms: conditions — Suicide; Accidental Injuries; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Using a parallel group design trial, our design considers the acceptability, feasibility and signals of impact of two different interventions: (1) the Family Safety Net for those whose household may benefit from lethal means reduction counseling due to having someone in their home who is struggling; and (2) a General Firearm Safety intervention for households with firearms who did not endorse an item on the family-focused mental health screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FSN Lethal Means Reduction (Experimental): * Participants will be screened into the lethal-means reduction-focused FSN program if they answer "yes" to one or more of the following questions:
  1. In the past two months, has anyone in your household been going through a rough time?
  2. In the past two months, has someone in your home seemed down, sad, or depressed?
  3. Are you worried that someone in your home is at risk of suicide?
  Participants are then assigned to either the MI FSN intervention or the Scripted FSN intervention
  Interventions: Behavioral: MI FSN - Lethal Means Reduction; Behavioral: Scripted FSN - Lethal Means Reduction
- General Firearm Safety Comparison (Active Comparator): General Firearm Safety
  * Participants will be screened into the general firearm safety arm of the program if they do not answer "yes" to any of the following questions:
  1. In the past two months, has anyone in your household been going through a rough time?
  2. In the past two months, has someone in your home seemed down, sad, or depressed?
  3. Are you worried that someone in your home is at risk of suicide?
  Participants are then assigned to either the General Firearm Safety Intervention or General Firearm Comparison
  Interventions: Behavioral: General Firearm Safety Intervention - General Firearm Safety; Behavioral: General Firearm Comparison - General Firearm Safety

INTERVENTIONS:
Behavioral: MI FSN - Lethal Means Reduction — Motivational Interviewing lethal means reduction, firearm storage supplies, Tailored text messages
  * Participate in a 15-20-minute motivational interviewing (MI) session conducted by trained University of Michigan research staff focused on encouraging suicide lethal means
  * Be offered to take home gun safety and lethal means reduction materials, including trigger locks, cable locks, ammo boxes, medication boxes and mental health resources
  * Receive 4 weeks of tailored text message reminders and encouragement
  Arms: FSN Lethal Means Reduction
Behavioral: Scripted FSN - Lethal Means Reduction — Scripted lethal means reduction, firearm storage supplies, tailored text messages
  * Participate in a 10-15-minute scripted session focused on gun safety and lethal means reduction
  * Be offered to home gun safety and lethal means reduction materials, including trigger locks, cable locks, ammo boxes, medication boxes and mental health resources
  * Receive 4 weeks of tailored text message reminders and encouragement
  Arms: FSN Lethal Means Reduction
Behavioral: General Firearm Safety Intervention - General Firearm Safety — General information on gun safety, firearm storage supplies, tailored text messages
  * Participate in a 10-minute scripted conversation about safe gun storage practice
  * Be offered to take home safe gun storage materials, including trigger locks, cable locks, and ammo boxes
  * Receive 4 weeks of tailored text message reminders and encouragement
  Arms: General Firearm Safety Comparison
Behavioral: General Firearm Comparison - General Firearm Safety — firearm storage supplies
  * Be offered to take home safe gun storage materials, including trigger locks, cable locks, and ammo boxes
  Arms: General Firearm Safety Comparison

SUMMARY:
Our parallel group clinical trial of the Family Safety Net (FSN) intervention addresses two main questions:

* Is the Family Safety Net (FSN) intervention feasible and acceptable in two formats: motivational interviewing (FSN MI) counseling session and scripted psychoeducational session (FSN Scripted), with a primarily Alaska Native population in Northwest Alaska?
* Secondarily, are there signals of efficacy at improving home safety (firearms unloaded, locked with ammunition separate) and dangerous medication locked?

All participants will complete a baseline survey with firearm storage questions as well as 3 questions about mental health concerns in their family (e.g. 'Are you worried that someone in your home is at risk of suicide?').

* If participants answer "yes" to any of these questions, they will be randomly assigned to one of the two FSN intervention groups (1 and 2 below).
* If they do not endorse any of the three family-focused mental health questions, they will be randomly assigned to one of two general firearm safety conditions (3 and 4 below).

  1. FSN MI group will participate in a 15-20-minute motivational interviewing (MI) session conducted by trained research staff focused on suicide lethal means reduction.
  2. FSN Scripted group will participate in a 10-minute scripted session focused on suicide lethal means reduction.

Both FSN groups (1 and 2):

* Can take home trigger locks, cable locks, ammo boxes, medication boxes and mental health resources
* Receive 4 weeks of tailored text message reminders and encouragement.
* Complete 1-month follow-up survey consisting of items related to firearm storage, and facilitating factors hypothesized to contribute to this behavior.
* Participants in both FSN conditions will be invited to participate in a semi-structured interview at follow-up focused on satisfaction and perceptions of the program.

  3 General gun safety intervention group will participate in a 10-minute scripted conversation about safe gun storage practice, and:
* Can take home trigger locks, cable locks, and ammo boxes.
* Receive 4 weeks of tailored text message reminders and encouragement.
* Complete 1-month follow-up survey consisting of items related to firearm storage, and facilitating factors hypothesized to contribute to this behavior.

  4. General gun safety comparison group:
* Can take home trigger locks, cable locks, and ammo boxes.
* Complete 1-month follow-up survey.

DETAILED DESCRIPTION:
The primary goal of this parallel-group clinical trial is to test the Family Safety Net (FSN) intervention in a primarily Alaska Native population in NW Alaska. The main question[s] it aims to answer are:

* Is the Family Safety Net (FSN) intervention acceptable in two formats, motivational interviewing counseling session, and scripted psychoeducational session, with a primarily Alaska Native population in Northwest Alaska?
* Secondarily, our small trial will describe signals of efficacy in improving home safe storage of firearms (unloaded, locked with ammunition separate from firearms) and medication.
* Participants will learn about the study from radio announcements or from receiving a respondent-driven sampling (RDS) coupon from another community member. We will aim to recruit an adult from at least 25% of the households in the community.
* Participants will be asked verbally if they qualify for the study, which will additionally be confirmed in the first few questions on the baseline survey, before they are consented. Participants qualify for the study if they:

  1. Are 18 or older
  2. Live in a home with at least one firearm
  3. Live in a home where young people (under 29) spend time
  4. Live in the region
  5. Are the only person from their household to participate in the study
  6. Have a cell phone that gets text messages
* If the participant qualifies and agrees to participate, they will be brought to a private room by the research staff. Research staff will walk through the screening criteria in the survey with the participant and go through the consent form on the iPad or on paper and answer the participant's questions. If they agree to participate, they will mark their consent, for both their participation and separately to have their session recorded, and additionally be offered a paper copy of the consent form to take home.
* Once consented, participants will be asked to complete a 10-15-minute baseline survey on the iPad. The survey will be done independently or with the help of the researcher if troubled by reading comprehension or navigating the iPad technology.
* Participants will be screened into either the lethal-means reduction-focused FSN program or the general firearm safety program based on their survey responses. If a respondent answers "yes" to one of the following questions, they are in the lethal-means reduction FSN arm of the program:

  1. In the past two months, has anyone in your household been going through a rough time?
  2. In the past two months, has someone in your home seemed down, sad, or depressed?
  3. Are you worried that someone in your home is at risk of suicide?

They are then randomly assigned into one of two groups using a grouped randomization table:

1. The lethal means reduction MI FSN group (n=10) will:

   1. Participate in a short 20-minute motivational interviewing (MI) session that includes:

      1. introduction to the session and setting the agenda;
      2. discussing the person's goals and strengths related to keeping loved ones safe through safe firearm and medication storage (e.g. making one's home safer to protect the youth or other family living there) and supporting wellness (i.e. mental health promotion);
      3. offering normative feedback about safe firearm storage practices within the community;
      4. talk about the benefits of safer firearm and medication storage practices (e.g. enhancing youth safety or avoiding youth harm);
      5. action planning to increase self-efficacy to overcome barriers and move toward reducing access to firearms and medications by locking and unloading all household guns and medications; and
      6. summarizing key content of the session to re-enforce benefits, goals, and values and support self-efficacy to facilitate safe firearm and medication storage practices and wellness support at home.
   2. Pick out safe storage devices to take home (e.g. trigger locks, cable locks, ammo boxes, medicine boxes, mental health crisis resources, local safety resources, etc.)
   3. Be told about the next steps of the study, including text messages, and follow-up survey and interview in about 4 weeks.
   4. Receive 4 weeks of text messages tailored by their survey responses (1x to 4x weekly depending on baseline survey responses). They may opt-out at any time.
2. The lethal means reduction bulleted script FSN group (n=10) will:

   1. Participate in a 15-minute conversation about lethal means reduction in their home, emphasizing that 10-minutes can save a life - the conversation includes discussing locations and storage of firearms, ammo, medications, and location of mental health crisis resources.
   2. Pick out safe storage devices to take home (e.g. trigger locks, cable locks, ammo boxes, medicine boxes, mental health crisis resources, local safety resources, etc.)
   3. Be told about the next steps of the study, including text messages, and follow-up survey and interview in about 4 weeks.
   4. Receive 4 weeks of text messages tailored by their survey responses (1x to 4x weekly depending on baseline survey responses). They may opt-out at any time.
3. The general firearm safety intervention group (n=10) will:

   1. Participate in a 10-minute conversation about safe firearm storage in their home including discussing locations and storage of firearms and ammo.
   2. Pick out safe storage devices to take home (e.g. trigger locks, cable locks, ammo boxes, local safety resources, etc.)
   3. Be told about the next steps of the study, including text messages, and follow-up survey and interview in about 4 weeks.
   4. Receive 4 weeks of text messages tailored by their survey responses (1x to 4x weekly depending on baseline survey responses). They may opt-out at any time.

   Researchers will compare people from the same population as the general gun safety group to see if household firearm storage practices change because of the scripted conversation around gun safety.
4. The general firearm safety comparison group (n=10) will:

   1. Pick out safe storage devices to take home (e.g. trigger locks, cable locks, ammo boxes, local safety resources, etc.)
   2. Be told about the next steps of the study, including a follow-up survey and interview in about 4 weeks.

All participants will be compensated for their time taking the baseline survey, regardless of group assignment.

* Participants will receive two RDS coupons at the end of their session to give to people in the community who they think would qualify and like to participate.
* The participants are instructed to check back in at the end of the day or later in the week to verify if either of the people they gave coupons to came in and participated.

One month after the initial session, a link will be sent to participants via text/email to complete a 10-15-minute (depending on skip logic) follow-up survey. The follow-up survey consists of items related to firearm storage and facilitating factors hypothesized to contribute to this behavior. The survey will include items focused on mechanisms of change, including self-efficacy, and on the current household gun storage (# and type of firearm; locked/unlocked, loaded/unloaded and location of ammo for each) and actions taken to support mental wellness for others in their home. Additionally, participants will also answer questions about their satisfaction with the FSN (acceptability, cultural responsiveness). For both comparison and intervention groups, the follow-up will capture a "snapshot" of current household firearm storage practices that day.

Participants will additionally be invited at the follow-up to take part in a 20-minute phone interview (semi-structured) also one month after their initial session. The follow-up semi-structured interview consists of questions about satisfaction with the program, what participants liked and didn't like, follow-up questions on the mental health concerns they have in their home, and follow-up on what they did with the home safety equipment they brought home and why as well as how the supplies worked for them.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18) who:

  * lives in the region,
  * Read and Understand English,
  * Live in a household with at least one gun,
  * Have a phone that can receive texts,
  * Lives in a household where young people (under 29) spend time

Exclusion Criteria:

* Someone else in the household has already participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of FSN | Through data collection, an average of 6 weeks
  The feasibility of the intervention will be tested by assessing the % of people who are eligible and agree (# agree/#eligible). The duration of each session will offer information about feasibility. We will also consider the level of attrition over the 4-week booster period, and the ability to collect follow-up data (target: 85% or 60 people) to assess participant satisfaction.
Acceptability of the intervention | Data collection for this aim will be done through data collection. Average 6 weeks
  Recorded FSN sessions will offer qualitative data about the acceptability of the intervention. Our analysis will capture instances within each session of acceptance through participants' willingness to discuss the connection between firearm or medication access and suicide risk; and curiosity or openness to learning about mental health resources. We will also make note of resistance (unacceptability), which likely include changes of subject, arguing and other 'avoidance talk'. We will consider the pattern of acceptability (and resistance) within each transcript. Across all FSN MI and script interventions, we will look for patterns of both acceptance and resistance to find trends in the data signaling the kinds of acceptable (and unacceptable) conversations within the FSN sessions.
Acceptability of the intervention | Through data collection. Average of 6 weeks
  FSN Follow-up Survey includes 4 items focused on participant satisfaction. Participants rank their favorite parts of the program and additionally, indicate with a 10 point Likert Scale, how much they agree with the following statements: (1) I am glad I participated in the Family Safety Net. (2) The Family Safety Net helped me meet my needs. (3) I would recommend Family Safety Net to a friend or family member. Answers will be aggregated for each item and overall. Items with an average 5.5 or more will be considered acceptable, and the intervention overall will be assessed by measurement average for all acceptability-related items of 5.5 or more.
Acceptability of the intervention | Through data collection. Average of 6 weeks
  FSN Follow-up Semi-Structured Interview includes 6 items focused on participant satisfaction. Participants are asked how each of the items they took home worked for them as well as the following questions: (1) What did you like best about the session? (2) Did you talk to anyone about your experience with FSN? (3) What did you think about the text messages you received? (4) Now that you did the whole Family Safety Net - the session a month ago, bringing home some safety supplies, and receiving text messages for the last month, what do you think is the best part of the program? (5) What might make it even better? (6) Is there anything else you want to tell us about your experience?

SECONDARY OUTCOMES:
Household Firearm Storage | Through data collection, an average of 6 weeks
  For each household firearm (up to five), the FSN Follow-up Survey asks them to characterize how that firearm is stored in their home today, indicating, "Yes", "No", or "Not Sure" for each home firearm. Questions for each firearm are: Is the firearm: (1) Stored in another's home for safety? (2) Locked with a cable or trigger lock? (3) In a locked gun safe/cabinet? (4) Unloaded? (5) Ammo stored away from the gun? (6) Ammo locked in an ammo box? (% baseline/% follow-up). We aim to answer how many (%) people went from storing firearms 'less safely' (e.g. unlocked) at baseline to more safely (e.g. locked) at follow-up, comparing results between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Wexler, PhD, MSW, Principal Investigator — University of Michigan
Locations (1):
- Maniilaq Association, Kotzebue, Alaska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone DM, Simon TR, Fowler KA, Kegler SR, Yuan K, Holland KM, Ivey-Stephenson AZ, Crosby AE. Vital Signs: Trends in State Suicide Rates - United States, 1999-2016 and Circumstances Contributing to Suicide - 27 States, 2015. MMWR Morb Mortal Wkly Rep. 2018 Jun 8;67(22):617-624. doi: 10.15585/mmwr.mm6722a1. PMID 29879094
- [Background] Blake I, Holck P, Provost EM. Alaska native mortality update: 2009-2013. Alsk Native Epidemiol. Published online 2016.
- [Background] Parker K. Alaska Trauma Registry. Trauma Admissions Involving Firearms; 2016.
- [Background] Anglemyer A, Horvath T, Rutherford G. The accessibility of firearms and risk for suicide and homicide victimization among household members: a systematic review and meta-analysis. Ann Intern Med. 2014 Jan 21;160(2):101-10. doi: 10.7326/M13-1301. PMID 24592495
- [Background] Horn A, Grossman DC, Jones W, Berger LR. Community based program to improve firearm storage practices in rural Alaska. Inj Prev. 2003 Sep;9(3):231-4. doi: 10.1136/ip.9.3.231. PMID 12966011
- [Background] Grossman DC, Stafford HA, Koepsell TD, Hill R, Retzer KD, Jones W. Improving firearm storage in Alaska native villages: a randomized trial of household gun cabinets. Am J Public Health. 2012 May;102 Suppl 2(Suppl 2):S291-7. doi: 10.2105/AJPH.2011.300421. Epub 2012 Mar 8. PMID 22401514
- [Background] Crosby AE, Ortega L, Stevens MR; Centers for Disease Control and Prevention (CDC). Suicides - United States, 2005-2009. MMWR Suppl. 2013 Nov 22;62(3):179-83. PMID 24264512
- [Background] Alaska bureau of vital statistics. Data and Statistics.; 2016.
- [Background] Collins PY, Delgado RA, Pringle BA, Roca C, Phillips A. Suicide prevention in Arctic Indigenous communities. Lancet Psychiatry. 2017 Feb;4(2):92-94. doi: 10.1016/S2215-0366(16)30349-2. No abstract available. PMID 28137384
- [Background] Yip PS, Caine E, Yousuf S, Chang SS, Wu KC, Chen YY. Means restriction for suicide prevention. Lancet. 2012 Jun 23;379(9834):2393-9. doi: 10.1016/S0140-6736(12)60521-2. PMID 22726520
- [Background] Zalsman G, Hawton K, Wasserman D, van Heeringen K, Arensman E, Sarchiapone M, Carli V, Hoschl C, Barzilay R, Balazs J, Purebl G, Kahn JP, Saiz PA, Lipsicas CB, Bobes J, Cozman D, Hegerl U, Zohar J. Suicide prevention strategies revisited: 10-year systematic review. Lancet Psychiatry. 2016 Jul;3(7):646-59. doi: 10.1016/S2215-0366(16)30030-X. Epub 2016 Jun 8. PMID 27289303
- [Background] van der Feltz-Cornelis CM, Sarchiapone M, Postuvan V, Volker D, Roskar S, Grum AT, Carli V, McDaid D, O'Connor R, Maxwell M, Ibelshauser A, Van Audenhove C, Scheerder G, Sisask M, Gusmao R, Hegerl U. Best practice elements of multilevel suicide prevention strategies: a review of systematic reviews. Crisis. 2011;32(6):319-33. doi: 10.1027/0227-5910/a000109. PMID 21945840
- [Background] Barber CW, Miller MJ. Reducing a suicidal person's access to lethal means of suicide: a research agenda. Am J Prev Med. 2014 Sep;47(3 Suppl 2):S264-72. doi: 10.1016/j.amepre.2014.05.028. PMID 25145749
- [Background] Strayer H, Craig J, Asay E, Haakenson A, Provost E. Alaska Native injury atlas: An update. In: Center IPPaANE, ed. 2014. Alaska Native Tribal Health Consortium; 2014.
- [Background] Ngo QM, Sigel E, Moon A, Stein SF, Massey LS, Rivara F, King C, Ilgen M, Cunningham R, Walton MA; FACTS Consortium. State of the science: a scoping review of primary prevention of firearm injuries among children and adolescents. J Behav Med. 2019 Aug;42(4):811-829. doi: 10.1007/s10865-019-00043-2. Epub 2019 Aug 1. PMID 31367940
- [Background] Wexler LM, Gone JP. Culturally responsive suicide prevention in indigenous communities: unexamined assumptions and new possibilities. Am J Public Health. 2012 May;102(5):800-6. doi: 10.2105/AJPH.2011.300432. Epub 2012 Mar 15. PMID 22420786
- [Background] Wexler L. Behavioral health services "Don't work for us": cultural incongruities in human service systems for Alaska Native communities. Am J Community Psychol. 2011 Mar;47(1-2):157-69. doi: 10.1007/s10464-010-9380-3. PMID 21052820
- [Background] Wexler L. Identifying colonial discourses in Inupiat young people's narratives as a way to understand the no future of Inupiat youth suicide. Am Indian Alsk Native Ment Health Res. 2009;16(1):1-24. doi: 10.5820/aian.1601.2009.1. PMID 19340763
- [Background] Wexler LM. Inupiat youth suicide and culture loss: Changing community conversations for prevention. Soc Sci Med. 2006 Dec;63(11):2938-48. doi: 10.1016/j.socscimed.2006.07.022. Epub 2006 Sep 6. PMID 16952416
- [Background] Philip J, Ford T, Henry D, Rasmus S, Allen J. Relationship of Social Network to Protective Factors in Suicide and Alcohol Use Disorder Intervention for Rural Yup'ik Alaska Native Youth. Interv Psicosoc. 2016 Apr;25(1):45-54. doi: 10.1016/j.psi.2015.08.002. Epub 2015 Oct 9. PMID 27110094
- [Background] Ullrich JS. For the love of our children: An indigenous connectedness framework. Altern Int J Indig Peoples. 2019;15(2):121.
- [Background] Allen J, Mohatt GV, Rasmus SM, et al. Cultural Interventions for American Indian and Alaska Native youth: The Elluam Tungiinun and Nagi Kicopi programs. In: Spicer P, Farrell P, Sarche M, Fitzgerald HE, eds. Child Psychology and Mental Health: Cultural and Ethno-Racial Perspectives, American Indian Child Psychology and Mental Health, Volume 2: Prevention and Treatment. Praeger Publishers; 2011.
- [Background] Burnette CE, Lesesne R, Temple C, Rodning CB. Family as the Conduit to Promote Indigenous Women and Men's Enculturation and Wellness: "I wish I had learned earlier". J Evid Based Soc Work (2019). 2020;17(1):1-23. doi: 10.1080/26408066.2019.1617213. Epub 2020 Jan 5. PMID 32133410
- [Background] Miller M, Azrael D, Barber C. Suicide mortality in the United States: the importance of attending to method in understanding population-level disparities in the burden of suicide. Annu Rev Public Health. 2012 Apr;33:393-408. doi: 10.1146/annurev-publhealth-031811-124636. Epub 2012 Jan 3. PMID 22224886
- [Background] Leavitt RA, Ertl A, Sheats K, Petrosky E, Ivey-Stephenson A, Fowler KA. Suicides Among American Indian/Alaska Natives - National Violent Death Reporting System, 18 States, 2003-2014. MMWR Morb Mortal Wkly Rep. 2018 Mar 2;67(8):237-242. doi: 10.15585/mmwr.mm6708a1. PMID 29494572
- [Background] Kegler SR, Stone DM, Holland KM. Trends in Suicide by Level of Urbanization - United States, 1999-2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 17;66(10):270-273. doi: 10.15585/mmwr.mm6610a2. PMID 28301448
- [Background] Ivey-Stephenson AZ, Crosby AE, Jack SPD, Haileyesus T, Kresnow-Sedacca MJ. Suicide Trends Among and Within Urbanization Levels by Sex, Race/Ethnicity, Age Group, and Mechanism of Death - United States, 2001-2015. MMWR Surveill Summ. 2017 Oct 6;66(18):1-16. doi: 10.15585/mmwr.ss6618a1. PMID 28981481
- [Background] Curtin SC, Warner M, Hedegaard H. Suicide Rates for Females and Males by Race and Ethnicity: United States.; 2016.
- [Background] Karch DL, Logan J, McDaniel D, Parks S, Patel N; Centers for Disease Control and Prevention (CDC). Surveillance for violent deaths--National Violent Death Reporting System, 16 states, 2009. MMWR Surveill Summ. 2012 Sep 14;61(6):1-43. PMID 22971797
- [Background] Brent DA. Firearms and suicide. Ann N Y Acad Sci. 2001 Apr;932:225-39; discussion; 239-40. doi: 10.1111/j.1749-6632.2001.tb05808.x. PMID 11411188
- [Background] Wexler L, Silveira ML, Bertone-Johnson E. Factors associated with Alaska Native fatal and nonfatal suicidal behaviors 2001-2009: trends and implications for prevention. Arch Suicide Res. 2012;16(4):273-86. doi: 10.1080/13811118.2013.722051. PMID 23137218
- [Background] Wolk CB, Jager-Hyman S, Marcus SC, Ahmedani BK, Zeber JE, Fein JA, Brown GK, Lieberman A, Beidas RS. Developing implementation strategies for firearm safety promotion in paediatric primary care for suicide prevention in two large US health systems: a study protocol for a mixed-methods implementation study. BMJ Open. 2017 Jun 24;7(6):e014407. doi: 10.1136/bmjopen-2016-014407. PMID 28647722
- [Background] Benjamin Wolk C, Van Pelt AE, Jager-Hyman S, Ahmedani BK, Zeber JE, Fein JA, Brown GK, Gregor CA, Lieberman A, Beidas RS. Stakeholder Perspectives on Implementing a Firearm Safety Intervention in Pediatric Primary Care as a Universal Suicide Prevention Strategy: A Qualitative Study. JAMA Netw Open. 2018 Nov 2;1(7):e185309. doi: 10.1001/jamanetworkopen.2018.5309. PMID 30646398
- [Background] Burch ES. Social Life in Northwest Alaska. University of Alaska Press; 2006.
- [Background] Craver A. Domestic function and Inupiaq households. Int J Circumpolar Health. 2004;Suppl 1:49-52. doi: 10.3402/ijch.v63i0.17775. PMID 15508467
- [Background] Heather N, Rollnick S, Bell A, Richmond R. Effects of brief counselling among male heavy drinkers identified on general hospital wards. Drug Alcohol Rev. 1996 Mar;15(1):29-38. doi: 10.1080/09595239600185641. PMID 16203349
- [Background] Resnicow K, Jackson A, Wang T, De AK, McCarty F, Dudley WN, Baranowski T. A motivational interviewing intervention to increase fruit and vegetable intake through Black churches: results of the Eat for Life trial. Am J Public Health. 2001 Oct;91(10):1686-93. doi: 10.2105/ajph.91.10.1686. PMID 11574336
- [Background] Rowhani-Rahbar A, Simonetti JA, Rivara FP. Effectiveness of Interventions to Promote Safe Firearm Storage. Epidemiol Rev. 2016;38(1):111-24. doi: 10.1093/epirev/mxv006. Epub 2016 Jan 13. PMID 26769724
- [Background] Silveira ML, Wexler L, Chamberlain J, Money K, Spencer RM, Reich NG, Bertone-Johnson ER. Seasonality of suicide behavior in Northwest Alaska: 1990-2009. Public Health. 2016 Aug;137:35-43. doi: 10.1016/j.puhe.2016.02.010. Epub 2016 Mar 24. PMID 27021788
- [Background] Miller M, Azrael D, Hemenway D. Household firearm ownership and suicide rates in the United States. Epidemiology. 2002 Sep;13(5):517-24. doi: 10.1097/00001648-200209000-00006. PMID 12192220
- [Background] Grossman DC, Mueller BA, Riedy C, Dowd MD, Villaveces A, Prodzinski J, Nakagawara J, Howard J, Thiersch N, Harruff R. Gun storage practices and risk of youth suicide and unintentional firearm injuries. JAMA. 2005 Feb 9;293(6):707-14. doi: 10.1001/jama.293.6.707. PMID 15701912
- [Background] Runyan CW, Brooks-Russell A, Betz ME. Points of Influence for Lethal Means Counseling and Safe Gun Storage Practices. J Public Health Manag Pract. 2019 Jan/Feb;25(1):86-89. doi: 10.1097/PHH.0000000000000801. No abstract available. PMID 29889177
- [Background] Bandura A. Self-Efficacy: The Exercise of Control. W.H. Freeman; 1997.
- [Background] Bandura A. Social Foundations of Thought and Action. Prentice-Hall; 1986.
- [Background] Carpenter CJ. A meta-analysis of the effectiveness of health belief model variables in predicting behavior. Health Commun. 2010 Dec;25(8):661-9. doi: 10.1080/10410236.2010.521906. PMID 21153982
- [Background] Grossman DC, Cummings P, Koepsell TD, Marshall J, D'Ambrosio L, Thompson RS, Mack C. Firearm safety counseling in primary care pediatrics: a randomized, controlled trial. Pediatrics. 2000 Jul;106(1 Pt 1):22-6. doi: 10.1542/peds.106.1.22. PMID 10878144
- [Background] Stevens MM, Olson AL, Gaffney CA, Tosteson TD, Mott LA, Starr P. A pediatric, practice-based, randomized trial of drinking and smoking prevention and bicycle helmet, gun, and seatbelt safety promotion. Pediatrics. 2002 Mar;109(3):490-7. doi: 10.1542/peds.109.3.490. PMID 11875146
- [Background] Kocalevent RD, Hinz A, Brahler E. Standardization of the depression screener patient health questionnaire (PHQ-9) in the general population. Gen Hosp Psychiatry. 2013 Sep-Oct;35(5):551-5. doi: 10.1016/j.genhosppsych.2013.04.006. Epub 2013 May 10. PMID 23664569
- [Background] Uebelacker LA, German NM, Gaudiano BA, Miller IW. Patient health questionnaire depression scale as a suicide screening instrument in depressed primary care patients: a cross-sectional study. Prim Care Companion CNS Disord. 2011;13(1):PCC.10m01027. doi: 10.4088/PCC.10m01027. PMID 21731830
- [Background] Rossom RC, Coleman KJ, Ahmedani BK, Beck A, Johnson E, Oliver M, Simon GE. Suicidal ideation reported on the PHQ9 and risk of suicidal behavior across age groups. J Affect Disord. 2017 Jun;215:77-84. doi: 10.1016/j.jad.2017.03.037. Epub 2017 Mar 16. PMID 28319695
- [Background] Wexler L, Moses J, Hopper K, Joule L, Garoutte J; LSC CIPA Team. Central role of relatedness in Alaska native youth resilience: Preliminary themes from one site of the Circumpolar Indigenous Pathways to Adulthood (CIPA) study. Am J Community Psychol. 2013 Dec;52(3-4):393-405. doi: 10.1007/s10464-013-9605-3. PMID 24185756
- [Background] Wexler L. Looking across three generations of Alaska Natives to explore how culture fosters indigenous resilience. Transcult Psychiatry. 2014 Feb;51(1):73-92. doi: 10.1177/1363461513497417. Epub 2013 Sep 6. PMID 24014514
- [Background] Trout L, Wexler L. Arctic Suicide, Social Medicine, and the Purview of Care in Global Mental Health. Health Hum Rights. 2020 Jun;22(1):77-89. PMID 32669791
- [Background] Lewis JP, Boyd K, Allen J, Rasmus S, Henderson T. "We Raise our Grandchildren as our Own:" Alaska Native Grandparents Raising Grandchildren in Southwest Alaska. J Cross Cult Gerontol. 2018 Sep;33(3):265-286. doi: 10.1007/s10823-018-9350-z. PMID 29797108
- [Background] Henderson TL, Dinh M, Morgan K, Lewis J. Alaska Native grandparents rearing grandchildren: A rural community story. J Fam Issues. 2017;38(4):547-572.
- [Background] Roy A, Noormohamed R, Henderson RI, Thurston WE. Promising healing practices for interventions addressing intergenerational trauma among Aboriginal youth: A scoping review. First Peoples Child Fam Rev. 2015;10(2):62-81.
- [Background] Ratcliff CL. Characterizing reactance in communication research: A review of conceptual and operational approaches. Commun Res. Published online 2019:0093650219872126.
- [Background] Gardner L, Leshner G. The Role of Narrative and Other-Referencing in Attenuating Psychological Reactance to Diabetes Self-Care Messages. Health Commun. 2016;31(6):738-51. doi: 10.1080/10410236.2014.993498. Epub 2015 Nov 3. PMID 26528578
- [Background] Firestone, R., Funaki, T., Dalhousie, S., Henry, A., Vano, M., Grey, J., Jull, A., Whittaker, R., Te Moringa, L. and Ni Mhurchu, C., 2018. Identifying and overcoming barriers to healthier lives.
- [Background] Vafeiadis M. The Role of Narratives, Frames and Visuals in Health Behavior Promotion: Increasing Public Awareness in the Era of Information Overload. Published online 2017.
- [Background] Alaska Department of Commerce Community and Economic Development. Community Information Summaries. Alsk Community Database. 2012. http://www.dced.state.ak.us/dca/commdb/CF_CIS.htm
- [Background] Pindus N, Kingsley T, Biess J, Levy D, Simington J, Hayes C. Housing needs of American Indians and Alaska Natives in Tribal areas: A report from the assessment of American Indian, Alaska Native, and Native Hawaiian housing needs: Executive summary. US Dep Hous Urban Dev Off Policy Dev Res. Published online 2017
- [Background] Hochbaum G, Rosenstock I, Kegels S. Health belief model. U S Public Health Serv. 1952;(Journal Article).
- [Background] Cummings KM, Jette AM, Rosenstock IM. Construct validation of the health belief model. Health Educ Monogr. 1978 Winter;6(4):394-405. doi: 10.1177/109019817800600406. PMID 299611
- [Background] Dillard JP, Shen L. On the nature of reactance and its role in persuasive health communication. Commun Monogr. 2005;72(2):144-168.
- [Background] Holmström É. Self-determination theory and the collaborative assessment and management of suicidality. Ment Health Rev J. 2020;25(1):75-83. doi:10.1108/MHRJ-09-2019-0029
- [Background] Kar Ray M, Wyder M, Crompton D, Kousoulis AA, Arensman E, Hafizi S, Van Bortel T, Lombardo C. PROTECT: Relational safety based suicide prevention training frameworks. Int J Ment Health Nurs. 2020 Jun;29(3):533-543. doi: 10.1111/inm.12685. Epub 2019 Dec 26. PMID 31880076
- [Background] Britton PC, Bryan CJ, Valenstein M. Motivational Interviewing for Means Restriction Counseling With Patients at Risk for Suicide. Cogn Behav Pract. 2016;23(1):51-61. doi:10.1016/j.cbpra.2014.09.004
- [Background] Ryan RM, Lynch MF, Vansteenkiste M, Deci EL. Motivation and Autonomy in Counseling, Psychotherapy, and Behavior Change: A Look at Theory and Practice 1ψ7. Couns Psychol. 2011;39(2):193-260. doi:10.1177/0011000009359313
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Preparing People for Change (2nd Ed.). Guilford Press; 2002. http://search.ebscohost.com/login.aspx?direct=true&db=psyh&AN=2002-02948-000&site=ehostlive
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Helping People Change. Guilford press; 2012.
- [Background] Jones SL, Jones PK, Katz J. Health belief model intervention to increase compliance with emergency department patients. Med Care. 1988 Dec;26(12):1172-84. doi: 10.1097/00005650-198812000-00007. PMID 3199913
- [Background] Jones CJ, Smith H, Llewellyn C. Evaluating the effectiveness of health belief model interventions in improving adherence: a systematic review. Health Psychol Rev. 2014;8(3):253-69. doi: 10.1080/17437199.2013.802623. Epub 2013 Jun 12. PMID 25053213
- [Background] Zak-Place J, Stern M. Health belief factors and dispositional optimism as predictors of STD and HIV preventive behavior. J Am Coll Health. 2004 Mar-Apr;52(5):229-36. doi: 10.3200/JACH.52.5.229-236. PMID 15029945
- [Background] Spoth R, Redmond C. Parent motivation to enroll in parenting skills programs: A model of family context and health belief predictors. J Fam Psychol. 1995;9(3):294-310. doi:10.1037/0893-3200.9.3.294
- [Background] Haas, Emily Joy. Toward harm reduction as a metatheory for health communication campaigns: An empirical study of harm reduction metatheory and the reconceptualized health belief model addressing motorcycle safety. PhD diss., Purdue University, 2012.
- [Background] Bulger EM, Kuhls DA, Campbell BT, Bonne S, Cunningham RM, Betz M, Dicker R, Ranney ML, Barsotti C, Hargarten S, Sakran JV, Rivara FP, James T, Lamis D, Timmerman G, Rogers SO, Choucair B, Stewart RM. Proceedings from the Medical Summit on Firearm Injury Prevention: A Public Health Approach to Reduce Death and Disability in the US. J Am Coll Surg. 2019 Oct;229(4):415-430.e12. doi: 10.1016/j.jamcollsurg.2019.05.018. Epub 2019 May 17. No abstract available. PMID 31108194
- [Background] Liu Y, Polman E, Liu Y, Jiao J. Choosing for others and its relation to information search. Organ Behav Hum Decis Process. 2018;147:65-75. doi:10.1016/j.obhdp.2018.05.005
- [Background] Oh H, Lee C. Culture and motivational interviewing. Patient Educ Couns. 2016 Nov;99(11):1914-1919. doi: 10.1016/j.pec.2016.06.010. Epub 2016 Jun 24. No abstract available. PMID 27401829
- [Background] Gayes LA, Steele RG. A meta-analysis of motivational interviewing interventions for pediatric health behavior change. J Consult Clin Psychol. 2014 Jun;82(3):521-35. doi: 10.1037/a0035917. Epub 2014 Feb 17. PMID 24547922
- [Background] Apodaca TR, Longabaugh R. Mechanisms of change in motivational interviewing: a review and preliminary evaluation of the evidence. Addiction. 2009 May;104(5):705-15. doi: 10.1111/j.1360-0443.2009.02527.x. PMID 19413785
- [Background] Rubak S, Sandbaek A, Lauritzen T, Christensen B. Motivational interviewing: a systematic review and meta-analysis. Br J Gen Pract. 2005 Apr;55(513):305-12. PMID 15826439
- [Background] Resnicow K, McMaster F. Motivational Interviewing: moving from why to how with autonomy support. Int J Behav Nutr Phys Act. 2012 Mar 2;9:19. doi: 10.1186/1479-5868-9-19. PMID 22385702
- [Background] Resnicow K, McMaster F, Rollnick S. Action reflections: a client-centered technique to bridge the WHY-HOW transition in Motivational Interviewing. Behav Cogn Psychother. 2012 Jul;40(4):474-80. doi: 10.1017/S1352465812000124. Epub 2012 Mar 14. PMID 22414686
- [Background] Miller WR, Rollnick S. Ten things that motivational interviewing is not. Behav Cogn Psychother. 2009 Mar;37(2):129-40. doi: 10.1017/S1352465809005128. PMID 19364414
- [Background] Butler CC, Rollnick S, Cohen D, Bachmann M, Russell I, Stott N. Motivational consulting versus brief advice for smokers in general practice: a randomized trial. Br J Gen Pract. 1999;49(445):611.
- [Background] Landro L. To Motivate Patients to Change, Doctors Stop Scolding. Wall Street Journal. April 29, 2013.
- [Background] Emmons KM, Rollnick S. Motivational interviewing in health care settings. Opportunities and limitations. Am J Prev Med. 2001 Jan;20(1):68-74. doi: 10.1016/s0749-3797(00)00254-3. PMID 11137778
- [Background] Israel, B. A., Eng, E., Schulz, A. J., & Parker, E. A. (2013). Introduction to methods for CBPR for health. Methods for community-based participatory research for health, 3-38.
- [Background] Wexler LM. Inupiat youth suicide: A critical ethnography of problem finding and response. 2005;Ph.D.
- [Background] Wexler L. Intergenerational dialogue exchange and action: Introducing a community-based participatory approach to connect youth, adults and elders in an Alaskan Native community. Int J Qual Methods. 2011;10(3):248-264.
- [Background] Barnett JD, Schmidt TC, Trainor B, Wexler L. A Pilot Evaluation of Culture Camps to Increase Alaska Native Youth Wellness. Health Promot Pract. 2020 May;21(3):363-371. doi: 10.1177/1524839918824078. Epub 2019 Feb 12. PMID 30755049
- [Background] Wexler L, Rataj S, Ivanich J, Plavin J, Mullany A, Moto R, Kirk T, Goldwater E, Johnson R, Dombrowski K. Community mobilization for rural suicide prevention: Process, learning and behavioral outcomes from Promoting Community Conversations About Research to End Suicide (PC CARES) in Northwest Alaska. Soc Sci Med. 2019 Jul;232:398-407. doi: 10.1016/j.socscimed.2019.05.028. Epub 2019 May 23. PMID 31151026
- [Background] Wexler L, Goodwin B. Youth and adult community member beliefs about Inupiat youth suicide and its prevention. Int J Circumpolar Health. 2006 Dec;65(5):448-58. doi: 10.3402/ijch.v65i5.18146. PMID 17319089
- [Background] Morgan DL. Focus Groups as Qualitative Research. SAGE Publications; 1996.
- [Background] King A, Simonetti J, Bennett E, Simeona C, Stanek L, Roxby AC, Rowhani-Rahbar A. Firearm storage practices in households with children: A survey of community-based firearm safety event participants. Prev Med. 2020 Feb;131:105952. doi: 10.1016/j.ypmed.2019.105952. Epub 2019 Dec 14. PMID 31843466
- [Background] Stott NC, Rollnick S, Rees MR, Pill RM. Innovation in clinical method: diabetes care and negotiating skills. Fam Pract. 1995 Dec;12(4):413-8. doi: 10.1093/fampra/12.4.413. PMID 8826057
- [Background] Velasquez MM, Hecht J, Quinn VP, Emmons KM, DiClemente CC, Dolan-Mullen P. Application of motivational interviewing to prenatal smoking cessation: training and implementation issues. Tob Control. 2000;9 Suppl 3(Suppl 3):III36-40. doi: 10.1136/tc.9.suppl_3.iii36. PMID 10982903
- [Background] Resnicow K, DiIorio C, Soet J, et al. Motivational Interviewing in medical and public health settings. In: Miller W, Rollnick S, eds. Motivational interviewing: Preparing people for change. 2nd ed. New York: Guildford Press; 2002:251-269.
- [Background] McMaster F, Resnicow K. Validation of the one pass measure for motivational interviewing competence. Patient Educ Couns. 2015 Apr;98(4):499-505. doi: 10.1016/j.pec.2014.12.014. Epub 2015 Jan 14. PMID 25624118
- [Background] Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med. 2007 Nov;22(11):1596-602. doi: 10.1007/s11606-007-0333-y. Epub 2007 Sep 14. PMID 17874169
- [Background] Dillard DA, Smith JJ, Ferucci ED, Lanier AP. Depression prevalence and associated factors among Alaska Native people: the Alaska education and research toward health (EARTH) study. J Affect Disord. 2012 Feb;136(3):1088-97. doi: 10.1016/j.jad.2011.10.042. Epub 2011 Dec 3. PMID 22138285
- [Background] Klaus NM, Mobilio A, King CA. Parent-adolescent agreement concerning adolescents' suicidal thoughts and behaviors. J Clin Child Adolesc Psychol. 2009 Mar;38(2):245-55. doi: 10.1080/15374410802698412. PMID 19283602
- [Background] De Los Reyes A, Augenstein TM, Wang M, Thomas SA, Drabick DAG, Burgers DE, Rabinowitz J. The validity of the multi-informant approach to assessing child and adolescent mental health. Psychol Bull. 2015 Jul;141(4):858-900. doi: 10.1037/a0038498. Epub 2015 Apr 27. PMID 25915035
- [Background] Simonetti JA, Rowhani-Rahbar A, King C, Bennett E, Rivara FP. Evaluation of a community-based safe firearm and ammunition storage intervention. Inj Prev. 2018 Jun;24(3):218-223. doi: 10.1136/injuryprev-2016-042292. Epub 2017 Jun 22. PMID 28642248
- [Background] Sobell LC, Sobell MB. Timeline Follow-Back. In: Litten RZ, Allen JP, eds. Measuring Alcohol Consumption: Psychosocial and Biochemical Methods. Humana Press; 1992:41-72. doi:10.1007/978-1- 4612-0357-5_3
- [Background] Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. BMJ. 2001 Nov 10;323(7321):1123-4. doi: 10.1136/bmj.323.7321.1123. No abstract available. PMID 11701584
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Background] Kelley K. Confidence Intervals for Standardized Effect Sizes: Theory, Application, and Implementation. J Stat Softw. 2007;20(8). doi:10.18637/jss.v020.i08
- [Background] Shenassa ED, Rogers ML, Spalding KL, Roberts MB. Safer storage of firearms at home and risk of suicide: a study of protective factors in a nationally representative sample. J Epidemiol Community Health. 2004 Oct;58(10):841-8. doi: 10.1136/jech.2003.017343. PMID 15365110
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] Shah S, Hoffman RE, Wake L, Marine WM. Adolescent suicide and household access to firearms in Colorado: results of a case-control study. J Adolesc Health. 2000 Mar;26(3):157-63. doi: 10.1016/s1054-139x(99)00064-6. PMID 10706163
- See also: Centers for Disease Control and Prevention, Web-based Injury Statistics Query and Reporting System (WISQARS). Fatal Injury Reports, Calculations were based on five years of most recently available data: 2013 to 2017. — https://www.cdc.gov/injury/wisqars